CLINICAL TRIAL: NCT05133908
Title: A Randomized Controlled Trial of Digital Cognitive Behavioral Therapy for Insomnia (dCBTi) for Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: dCBTi for Adults With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Wai Sze, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA210505
Record Dates: First submitted 2021-11-22; First posted 2021-11-24 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Insomnia
Keywords: Digital intervention; Cognitive Behavioral Therapy for Insomnia; Treatment efficacy; Treatment adherence
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All outcome measures will be administered via online surveys
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Sleep Hygiene and Self-Monitoring Control (Active Comparator): Participants assigned to this condition will receive an app to track sleep and offers sleep hygiene recommendations
  Interventions: Behavioral: Sleep Hygiene and Self-Monitoring Control
- dCBTi-ADHD (Experimental): Participants assigned to this condition will receive a 7-module digital cognitive behavioral therapy for insomnia (dCBTi) tailored for adults with ADHD
  Interventions: Behavioral: dCBTi-ADHD

INTERVENTIONS:
Behavioral: Sleep Hygiene and Self-Monitoring Control — An app with self-monitoring function and videos and written materials about sleep hygiene will be provided.
  Arms: Digital Sleep Hygiene and Self-Monitoring Control
Behavioral: dCBTi-ADHD — The dCBTi adopts a multi-module approach, consisting of 7 weekly modules including psychoeducation on sleep and ADHD, insomnia, organization strategies and distractibility reduction skills, sleep hygiene, sleep restriction and prescription, circadian-related activity scheduling, stimulus control, relaxation and worry time, cognitive restructuring, and relapse prevention. In each module, participants will watch short videos to learn strategies to improve their sleep. A virtual coach is also included in the app functionality. It will be in the form of a text-based forced-choice conversation bot. It will initiate conversations with the users to check their understanding of treatment materials and guide them to come up with specific action plans to implement the treatment strategies.
  Arms: dCBTi-ADHD

SUMMARY:
The current study aims to evaluate the efficacy and feasibility of a digital application-based CBTi treatment devised for adults with ADHD and insomnia compared to self-monitoring and sleep hygiene control condition.

DETAILED DESCRIPTION:
Participants would be randomly assigned to the experimental or sleep diary self-monitoring (control) group. Participants in the experimental group would use a digital application for seven weeks, whereas participants in the control group would watch psychoeducation videos on sleep hygiene and enter sleep diary measures using the application for seven weeks.

Question 1:

Does dCBTi work better than the active control?

Hypothesis 1:

Improvement in insomnia (immediately after treatment and at 1-month follow-up) would be greater for the experimental group than the active control group.

Question 2:

Does improvement in insomnia due to dCBTi lead to improvement in ADHD outcomes?

Hypothesis 2:

Improvement in ADHD outcomes would be greater for the experimental group than the active control group. The effect of dCBTi on ADHD outcomes would be mediated by improvement in insomnia.

Question 3:

Does improvement in insomnia due to dCBTi lead to improvement in mental well-being?

Hypothesis 3:

Improvement in outcomes related to mental well-being would be greater for the experimental group than the active control group. The effect of dCBTi on outcomes related to mental well-being would be mediated by improvement in insomnia.

ELIGIBILITY:
Inclusion Criteria:

* (a) Hong Kong resident,
* (b) Aged between 18-60,
* (c) Diagnosed with ADHD,
* (d) Able to read and write Chinese,
* (e) Has regular access to a smart phone and internet,
* (f) Insomnia severity index ⩾10

Exclusion Criteria:

* (a) Having comorbid bipolar disorder, psychosis, suicidality, moderately severe to severe depression, narcolepsy, and/or hypersomnolence disorder,
* (b) Having medical conditions that might affect sleep (e.g., serious physical concerns necessitating surgery, risk of falls, epilepsy),
* (c) Having night shift schedules at work,
* (d) Currently receiving psychological intervention for insomnia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Insomnia Severity Index (ISI) | 13 weeks from baseline
  Insomnia symptoms measured by the Insomnia Severity Index (ISI). The score ranges from 0 to 24. Higher scores indicate greater levels of insomnia symptoms

SECONDARY OUTCOMES:
Changes in total sleep time (TST) | 13 weeks from baseline
  Total sleep time (TST) measured by Consensus Sleep Diary. Its units is minutes. Higher TST indicates longer total sleep duration.
Changes in sleep efficiency (SE) | 13 weeks from baseline
  Sleep efficiency (SE) measured by Consensus Sleep Diary. It ranges from 0 to 100%, the higher indicates better sleep
Changes in sleep onset latency (SOL) | 13 weeks from baseline
  Sleep onset latency (SOL) measured by Consensus Sleep Diary. Its unit is minutes. Longer SOL indicates greater levels of insomnia
Changes in midsleep time (MST) | 13 weeks from baseline
  Midsleep time (MST) measured by Consensus Sleep Diary. Its unit is time. Earlier MST indicates earlier overall timing of sleep.
Changes in fatigue | 13 weeks from baseline
  Fatigue measured by the Fatigue Assessment Scale (FAS). The score ranges from 10 to 50, the higher the greater levels of fatigue
Changes in depressive symptoms | 13 weeks from baseline
  Depressive symptoms measured by the Patient Health Questionnaire - 9 (PHQ-9). The score ranges from 0 to 27, the higher the more depressed
Changes in anxiety symptoms | 13 weeks from baseline
  Anxiety symptoms measured by the Generalized Anxiety Disorder 7-item Scale (GAD-7). The score ranges from 0 to 21, the higher the more anxious
Changes in mental wellbeing | 13 weeks from baseline
  Mental well-being measured by the Warwick Edinburgh Mental Well-being Scale (WEMWBS). The score ranges from 14 to 70, the higher the greater level of mental well-being
Changes in ADHD symptoms | 13 weeks from baseline
  ADHD symptoms measured by the Adult ADHD Self-Report Scale (ASRS). The score ranges from 0 to 72, the higher the greater symptom severity
Changes in functional impairment due to ADHD symptoms | 13 weeks from baseline
  Functional impairment due to ADHD symptoms measured by three questions evaluating the extent to which individuals' ADHD symptoms affect their ability to function in the domains of work/study, housekeeping, and social relationships. The questions are rated on a 4-point scale, with higher ratings indicating higher level of impairment
Changes in executive skills | 13 weeks from baseline
  Executive skills measured by the Executive Skills Questionnaire-Revised (ESQ-R). The score ranges from 0 to 75, the lower the stronger executive skills

CONTACTS AND LOCATIONS:
Overall Officials: Wai Sze Chan, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available for sharing with other researchers for secondary analysis upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From after the study findings have been published to 5 years afterwards.
Access Criteria: The request party has a pre-registration of the research that requires data from the present study indicating clearly what data are required and other criteria as the PI deem appropriate.